CLINICAL TRIAL: NCT06814431
Title: Study on the Incidence of Malignant Neoplasms in Patients with Parkinson's Disease and Heterozygous Mutation of the GBA Gene
Acronym: ONCOGBA
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 133/2023/OSS/AUSLRE
Record Dates: First submitted 2025-01-29; First posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Parkinson's Disease (PD)
Keywords: Parkinson's Disease; Neoplasms; GBA1; Genetic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GBA-PD Cohort: Parkinson's disease (PD) patients diagnosed based on the "United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria". Patients in this group must have a documented heterozygous pathogenic variant in the GBA1 gene.
- Idiopathic PD Cohort: This cohort includes patients diagnosed with Parkinson's disease (PD) based on the "United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria". Patients in this group do not have any documented heterozygous pathogenic variants in the GBA1 or LRRK2 genes.

SUMMARY:
This multicenter retrospective observational study investigates the incidence of malignant neoplasms in Parkinson's disease (PD) patients carrying heterozygous pathogenic variants in the GBA1 gene. The study compares these patients to individuals with idiopathic PD and to the general population within a large national cohort.

The rationale for the study lies in the growing evidence indicating an increased risk of malignant neoplasms in patients affected by Gaucher disease.

The primary objective is to assess whether PD patients with GBA1 mutations have a higher incidence of malignant neoplasms compared to the general population. Secondary objectives include comparing the incidence of malignant neoplasms between GBA1-PD and idiopathic PD patients, as well as between idiopathic PD patients and the general population. Additionally, the study aims to characterize oncological conditions by sex, age, center, and tumor site, with specific attention to distinguishing hematologic tumors from solid tumors.

By identifying potential associations between GBA1 mutations and malignancies in PD, the findings could guide more comprehensive patient management, including screening for malignant neoplasms alongside Parkinson's disease care.

DETAILED DESCRIPTION:
The study will involve a network composed by different Italian Movement Disorders Centres and the corresponding local cancer registries, responsible for the active collection of cancer cases. Data will be collected from approximately 3000 consecutive Parkinson's disease (PD) patients, including about 500 patients carrying GBA1 mutations and 2500 idiopathic PD. Data about the presence of malignancies will be extracted from the Local Cancer Registries for each patient.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Diagnosis of Parkinson's Disease through the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria for Parkinson's Disease.

Exclusion Criteria:

* Uncertain diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from a network of Italian neurology centers with extensive experience in studying GBA-associated PD, in collaboration with local cancer registries. The study will include approximately 3,000 consecutive PD patients, subdivided into 500 patients with GBA mutations and 2,500 patients with idiopathic PD.
  These participants will be compared with data from cancer registries to investigate potential associations between GBA mutations and malignancies. The population is drawn from specialized movement disorder centers and represents a clinically well-characterized cohort with access to standardized diagnostic and follow-up procedures.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Increased Incidence of Malignant Neoplasms in Parkinson's Disease Patients with GBA1 Mutation Compared to the General Population | From birth to a maximum of 36 months after enrollment
  The incidence of malignant neoplasms in Parkinson's disease (PD) patients carrying the GBA1 mutation (GBA1-PD) will be calculated and compared to that of the general population to assess any potential increase in risk.

SECONDARY OUTCOMES:
Evaluation of Increased Incidence of Malignant Neoplasms in Parkinson's Disease Patients with GBA1 Mutation Compared to Non-Genetic Parkinson's Disease Patients | From birth to a maximum of 36 months after enrollment
  The incidence of malignant neoplasms in Parkinson's disease (PD) patients carrying the GBA1 mutation (GBA1-PD) will be compared to that of idiopathic PD patients using a Chi-Square test to evaluate statistical significance
Evaluation of Increased Incidence of Malignant Neoplasms in Idiopathic Parkinson's Disease Patients Compared to the General Population | From birth to a maximum of 36 months after enrollment
  The incidence of neoplasms in patients with idiopathic Parkinson's disease (PD) will be compared to that of the general population.
Description of Oncological Condition Incidence by Sex, Age, Center, and Tumor Site, with Specific Focus on Hematologic Versus Solid Tumors | From birth to a maximum of 36 months after enrollment
  Logistic regression analysis will be conducted to evaluate the association between neoplasms and PD subgroups (GBA1 and idiopathic PD), accounting for clinical and demographic covariates.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Ospedale A. Perrino, Brindisi
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia
  - Ospedale Santa Chiara di Trento, Trento

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stirnemann J, Belmatoug N, Camou F, Serratrice C, Froissart R, Caillaud C, Levade T, Astudillo L, Serratrice J, Brassier A, Rose C, Billette de Villemeur T, Berger MG. A Review of Gaucher Disease Pathophysiology, Clinical Presentation and Treatments. Int J Mol Sci. 2017 Feb 17;18(2):441. doi: 10.3390/ijms18020441. PMID 28218669
- [Background] Mistry PK, Taddei T, vom Dahl S, Rosenbloom BE. Gaucher disease and malignancy: a model for cancer pathogenesis in an inborn error of metabolism. Crit Rev Oncog. 2013;18(3):235-46. doi: 10.1615/critrevoncog.2013006145. PMID 23510066